CLINICAL TRIAL: NCT00360009
Title: Cognition and Mood in Parkinson's Disease (PD) in Subthalamic Nucleus (STN) Versus Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Brief Title: Effects of Deep Brain Stimulation on Motor, Mood, and Cognitive Symptoms in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 303-2002; K23NS044997 (NIH)
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Parkinson disease; PD; deep brain stimulation; DBS; subthalamic nucleus; STN; globus pallidus interna; GPi; mood; motor symptoms; cognition; emotion; memory; attention; tremor; rigidity; bradykinesia
MeSH Terms: conditions — Parkinson Disease; Tremor; Muscle Rigidity; Hypokinesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- STN DBS (Active Comparator): Patients who underwent deep brain stimulation (DBS) of the subthalamic nucleus (STN) to treat Parkinson's disease (PD)
  Interventions: Procedure: DBS of the STN
- GPI DBS (Active Comparator): Patients who underwent deep brain stimulation (DBS) of the globus pallidus interna (GPi) to treat Parkinson's disease (PD)
  Interventions: Procedure: DBS of the GPI
- no DBS (No Intervention): non-DBS PD patient control group

INTERVENTIONS:
Procedure: DBS of the STN — Patients undergo Deep Brain Stimulation (DBS) of the subthalamic nucleus (STN) to treat Parkinson's Disease, using a Medtronic 3387 device.
  Arms: STN DBS
Procedure: DBS of the GPI — Patients undergo Deep Brain Stimulation (DBS) of the globus pallidus interna (Gpi) to treat Parkinson's disease, using a Medtronic 3387 device.
  Arms: GPI DBS

SUMMARY:
The purpose of this trial is to study the mood and cognitive effects of deep brain stimulation in Parkinson's disease.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) of the subthalamic nucleus (STN) and the globus pallidus interna (GPi) has been shown to relieve the motor symptoms of Parkinson's disease (PD) such as tremor, rigidity, and bradykinesia. However, there is increasing evidence that DBS may be associated with a significant number of mood and cognitive changes.

The aims of this study are to characterize and compare the mood and cognitive effects associated with DBS of the STN and GPi, to delineate regions within or around the STN and GPi that are associated with specific mood and cognitive changes when DBS is applied to these areas, and to assess the relative effectiveness of right versus left STN or GPi stimulation on mood and cognition.

In the study, researchers will compare motor, mood, and cognitive function in people with PD who have had DBS treatment with control subjects (or individuals with PD who have not had DBS). The scientists will characterize the types and incidence of mood and cognitive changes that occur during DBS in each target (STN and GPi), compare the targets, and examine the role of lead location.

The study will enroll 62 participants-10 control subjects (individuals with PD who have not had DBS), and 52 individuals with PD who are scheduled for DBS; the site of the implant (STN or GPi) will be randomly assigned. Participants will perform motor, mood, and cognitive tests (following 6 months of stimulation) over a 2-day period. Duration of the trial for participants is 6 months and includes a 2-night hospital stay.

Findings from this study may help researchers better understand how DBS affects non-motor circuitry.

ELIGIBILITY:
Inclusion Criteria:

* Intractable, disabling PD with motor fluctuations, dyskinesias, or freezing episodes
* Age between 30-75 years
* Unsatisfactory clinical response to maximal medical management (with trials of both higher and lower doses of anti-Parkinsonian drugs)
* A stable and optimal medical regimen of anti-Parkinsonian drug therapy for at least three months prior to surgery
* Patients must be right-handed to be included in the study since mood and cognition are being analyzed and right hemisphere dominant patients could confound the results.

Exclusion Criteria:

* Clinically significant medical disease that would increase risk of developing pre- or postoperative complications (e.g., significant cardiac or pulmonary disease, uncontrolled hypertension)
* Evidence of secondary or atypical parkinsonism as suggested by the presence of any of the following: 1) history of stroke(s), 2) exposure to toxins or neuroleptics, 3) history of encephalitis, 4) neurological signs of upper motor neuron disease, cerebellar involvement, supranuclear gaze palsy, or significant orthostatic hypotension
* MRI scan with significant evidence of brain atrophy or other abnormalities (e.g., lacunar infarcts or iron deposits in the putamen)
* The Mattis Dementia Rating Scale will be used to assess the level of intellectual function and patients will be excluded with scores reflecting clinical dementia
* A major psychiatric disorder on the Structured Clinical Interview for DSM-IV (SCID-IV).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Okun, MD, Principal Investigator — University of Florida; Kelly Foote, MD, Principal Investigator — University of Florida; Hubert Fernandez, MD, Principal Investigator — University of Florida; Ramon Rodriguez, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida College of Medicine, Department of Neurology, McKnight Brain Institute, 100 South Newell Drive, L-3 100, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- No Deep Brain Stimuation (DBS) Control Group: A control group of PD patients that have not undergone surgical intervention (ie. DBS).
- Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS): Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) intervention to treat Parkinson's disease (PD)
- Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS): Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS) intervention to treat Parkinson's Disease (PD)
Period: Overall Study
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Started | 10 | 26 | 26
Completed | 10 | 22 | 23
Not Completed | 0 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS) | Total
Number analyzed (Participants) | 10 | 26 | 26 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 16 | 19 | 40
  >=65 years | 5 | 10 | 7 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 8 | 20
  Male | 6 | 18 | 18 | 42
Region of Enrollment [Number; unit: participants]
  United States | 10 | 26 | 26 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean T-score of Visual Analogue Mood Scales (VAMS) Angry State
Description: VAMS measure mood states using scales that have a neutral face/word at the top of a vertical line and a specific mood face/word at the bottom of the line. Respondents indicate a point on the line that describes how they are feeling and a raw score between 0-100 is obtained. The raw score is converted to a T-score. The mean pre and post-DBS T-scores are compared. A negative difference in T-score(-0.5) indicates a reduction in mood from pre to post-DBS while a positive T-score difference(2.4) denotes an increase in mood. The larger the absolute T-score value, the greater the mean change in mood.
Time Frame: Pre-surgery baseline to 6 months of DBS stimulation
Population: Control Group data not reported for this outcome measure because the purpose of the Control Group was just to test effects of fatigue.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 0 | 22 | 23
T-score |  | 5.3 (10.2) | -0.1 (5.3)

2. Secondary Outcome: Change in Spielberger State-Trait Anxiety Inventory (STAI)
Description: STAI measures anxiety. The questionnaire asks the patients how they feel and allows them to respond on a frequency scale that ranges from 1(not at all) to 4(almost always/very much so). Scores range from 20-80 and the higher the score the greater the anxiety level. The raw score is converted to a T-score. The mean pre and post-DBS T-scores are compared. A negative difference in T-score(-1.4) indicates a reduction in anxiety from pre to post-DBS while a positive T-score difference (0.4) denotes an increase in anxiety. The larger the absolute T-score value,the greater the mean change in anxiety.
Time Frame: Pre-surgery baseline to 6 months of DBS stimulation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 0 | 22 | 23
T-score |  | -3.3 (13.4) | 0.3 (13.6)

3. Secondary Outcome: Change in Beck Depression Inventory (BDI)
Description: BDI is a questionnaire used to measure depression. There is a four-point scale for each of the 21-items of the questionnaire with scores ranging from 0 to 3. Total raw scores range from 0 to 63. The higher the score the greater the severity of depression. The raw score is converted to a T-score. The mean pre and post-DBS T-scores are compared. A negative difference in T-score(-3.7) indicates a reduction in depression from pre to post-DBS while a positive T-score difference (0.4) denotes an increase in depression. The larger the absolute T-score value,the greater the mean change in depression.
Time Frame: Pre-surgery baseline to 6 months of DBS stimulation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 0 | 22 | 23
T-score |  | -2.8 (6.3) | -4.6 (5.4)

4. Secondary Outcome: Change in Letter Fluency Tasks (LFT)
Description: LFT assess frontal lobe function. Performance measure is number of words beginning with a specific letter generated in 1 min. Although no range of possible scores,the more words named in allotted time,the higher the predicted frontal lobe function. Raw score is converted to T-score. The mean pre and post-DBS T-scores are compared. A negative difference in T-score(-2.6) signifies a reduction in task performance from pre to post-DBS while a positive T-score difference(0.7) denotes an increase in task performance. The larger the absolute T-score value,the greater the mean change in performance.
Time Frame: Pre-surgery baseline to 6 months of DBS stimulation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 0 | 22 | 23
T-score |  | -5.6 (6.7) | 0.3 (10.7)

5. Primary Outcome: Change in Visual Analogue Mood Scales (VAMS) Afraid State
Description: as for outcome 1
Time Frame: Pre-surgery baseline to 6 months of DBS stimulation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 0 | 22 | 23
T-score |  | 1.3 (16.9) | -2.2 (13.0)

6. Primary Outcome: Change in Visual Analogue Mood Scales (VAMS) Confused State
Description: as for outcome 1
Time Frame: Pre-surgery baseline to 6 months of DBS stimulation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 0 | 22 | 23
T-score |  | 5.7 (15.4) | 1.3 (11.0)

7. Primary Outcome: Change in Visual Analogue Mood Scales (VAMS) Energetic State
Description: as for outcome 1
Time Frame: Pre-surgery baseline to 6 months of DBS stimulation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 0 | 22 | 23
T-score |  | -1.4 (12.3) | 2.0 (18.7)

8. Primary Outcome: Change in Visual Analogue Mood Scales (VAMS) Happy State
Description: as for outcome 1
Time Frame: Pre-surgery baseline to 6 months of DBS stimulation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 0 | 22 | 23
T-score |  | 2.9 (17.2) | 5.0 (13.8)

9. Primary Outcome: Change in Visual Analogue Mood Scales (VAMS) Sad State
Description: as for outcome 1
Time Frame: Pre-surgery baseline to 6 months of DBS stimulation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 0 | 22 | 23
T-score |  | -2.4 (17.8) | -1.0 (13.0)

10. Primary Outcome: Change in Visual Analogue Mood Scales (VAMS) Tense State
Description: as for outcome 1
Time Frame: Pre-surgery baseline to 6 months of DBS stimulation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 0 | 22 | 23
T-score |  | -2.0 (17.5) | -8.5 (20.0)

11. Primary Outcome: Change in Visual Analogue Mood Scales (VAMS) Tired State
Description: as for outcome 1
Time Frame: Pre-surgery baseline to 6 months of DBS stimulation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 0 | 22 | 23
T-score |  | -8.5 (12.0) | -2.0 (13.5)

ADVERSE EVENTS:
Arm/Group | No Deep Brain Stimuation (DBS) Control Group | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS)
Serious Adverse Events (participants affected / at risk) | 0/10 | 6/26 | 8/26
Other Adverse Events (participants affected / at risk) | 0/10 | 25/26 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Deep Brain Stimuation (DBS) Control Group (N=10) | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) (N=26) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS) (N=26)
Confusion/Disorientation/Difficulty Concentrating/Distractability (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia Resulting in Death (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Symptomatic Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Symptomatic Venous Hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Air Embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety/Feafulness/Preocupation with Health (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage Resulting in Death (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Deep Brain Stimuation (DBS) Control Group (N=10) | Subthalamic Nucleus (STN) Deep Brain Stimulation (DBS) (N=26) | Globus Pallidus Interna (GPi) Deep Brain Stimulation (DBS) (N=26)
Depression/Tearful/Decreased Confidence/Loss of Motivation/Feelings of Guilt (Psychiatric disorders) | 0 (0) | 20 (20) | 7 (7)
Anxiety/Fearfulness/Preoccupation with Health (Psychiatric disorders) | 0 (0) | 14 (14) | 6 (6)
Difficulty with Speech and Language/Increased Speech (Nervous system disorders) | 0 (0) | 8 (8) | 10 (10)
Confusion/Disorientation/Difficulty Concentrating/Distractibility (Psychiatric disorders) | 0 (0) | 7 (7) | 4 (4)
Irritability/Disruptive of Aggressive Behavior (Psychiatric disorders) | 0 (0) | 10 (10) | 5 (5)
Obsessive-Compulsive Tendencies (Psychiatric disorders) | 0 (0) | 5 (5) | 2 (2)
Manic Tendencies (Psychiatric disorders) | 0 (0) | 5 (5) | 1 (1)
Worsening of Memory (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3)
Sleep Disturbance/Vivid Dreaming/Increased Somnolence (Nervous system disorders) | 0 (0) | 14 (14) | 11 (11)
Fatigue/Tired (General disorders) | 0 (0) | 11 (11) | 3 (3)
Pain (General disorders) | 0 (0) | 9 (9) | 2 (2)
Worsening of Balance/Gait Disturbance/Freezing (Nervous system disorders) | 0 (0) | 6 (6) | 5 (5)
Decreased Libido (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 5 (5)
Dizziness/Lightheadedness/Orthostasis (General disorders) | 0 (0) | 4 (4) | 2 (2)
Weakness (General disorders) | 0 (0) | 4 (4) | 1 (1)
Weight Loss (General disorders) | 0 (0) | 3 (3) | 2 (2)
Headache/Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3)
Difficulty with Urination/Urinary Urgency/Distended Bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Anorexia (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3)
Pain/Discomfort/Pruritus/Erythema at Sight of Incision (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Stomach Cramps/Constipation/Indegestion (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Cold/Low-grade Fever (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Dry Mouth (General disorders) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No